CLINICAL TRIAL: NCT04318054
Title: Medical Benefit Evaluation of Ambulatory Activity Combining Rehabilitation and Therapeutic Education, Using an Intelligent Electric Bike for the Health, for the Effort Rehabilitation and the Quality of Life Improvement for Patients Suffering of Moderate Fibromyalgia.
Brief Title: Medical Benefit Evaluation of Ambulatory Activity Combining Rehabilitation and Therapeutic Education, Using an Intelligent Electric Bike for the Health, for the Effort Rehabilitation and the Quality of Life Improvement for Patients Suffering of Moderate Fibromyalgia (FIBROVELIS)
Acronym: Fibrovelis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC19.128
Record Dates: First submitted 2020-01-24; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Fibromyalgia; Chronic Pain; Adapted Physical Activity; Therapeutic Education; Electric Bike
Keywords: fibromyalgia; chronic pain; adapted physical activity; therapeutic education; electric bike
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Immediate intervention group : fibromyalgia patients consulting in Grenoble Alps University Hospital who will practice, in the 2 months following the randomization, an ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health during 8 weeks (2 times by week).
  Deferred intervention group : fibromyalgia patients consulting in Grenoble Alps University Hospital who will practice, one year after the inclusion, an ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health during 8 weeks (2 times by week).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention group (Experimental): fibromyalgia patients consulting in Grenoble Alps University Hospital who will practice, in the 2 months following the randomization, an ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health during 8 weeks (2 times by week).
  Interventions: Other: Ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health.
- Deferred intervention group (Other): Deferred intervention group : fibromyalgia patients consulting in Grenoble Alps University Hospital who will practice, one year after the inclusion, an ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health during 8 weeks (2 times by week).
  Interventions: Other: Ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health.

INTERVENTIONS:
Other: Ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health. — fibromyalgia patients consulting in Grenoble Alps University Hospital who will practice an ambulatory activity combining rehabilitation and therapeutic education, using an Intelligent Electric Bike for the Health during 8 weeks (2 times by week).

SUMMARY:
The aim of this study is to decrease the impact of the fibromyalgia on the daily quality of life of the patients suffering of moderate fibromyalgia at 6 months by the practice of an adapted physical activity coupled with therapeutic education workshop.

DETAILED DESCRIPTION:
Fibromyalgia is chronic pain syndrome expressed as fluctuacting musculotendinous or articular pain and chronic tiredness. Among the non-pharmacological treatments, apart the "psychological" accompanying, the EULAR (European League Against Reumatism) recommends the physical activity in first intention. Thus, physical reconditioning has an important place in fibromyalgia. Aerobic conditioning or reconditioning programs for effort induce for some patients a benefit on quality of life, tiredness and pain. In France, these programmes are mostly carried out in "follow-up and rehabilitation" type care structures.

Outdoor exercise re-training with the Intelligent Electric Bike for Health combined with therapeutic education sessions are proposed in the study. These activities, adapted to each group and patient, can best achieve the objective in an ambulatory format closer to the patient's daily life.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Patient available for a following of 18 months
* Patient available for go to sessions of Intelligent Electric Bike for the Health, 2 half-day by week during 8 weeks in the 2 months following the randomization.
* confirmed fibromyalgia according to the criteria of the American College of Rhumatology 2010 since at least one year with a stable treatment since at least 3 months.
* Patients with a score of 39 ≤ FIQ < 59 (moderate fibromyalgia impact)
* Patient in capacity to pedal on a bike outside.
* Patient who haven't contraindications at the practice of an moderate physical activity or bike (acute coronary pathology less than 2 years, locomotor problems of the spine or lower limbs incompatible with the bike practice).
* Weight lower than 125 kg (maximal load for the Intelligent Electric Bike for the Health).
* Patient having signed the written consent after appropriate information and delivery of the information note.
* Patient affiliated at the social security or beneficiary of such a scheme

Exclusion Criteria:

* Substantial variation of the therapeutic care in the 3 months previous the inclusion (change of drug class, beginning of physical reconditioning in an unit of follow-up and rehabilitation care, or a cognitive-behavioral technique)
* Patient with treatement which can deteriorate the attention
* Patient suffering of a serious chronic desease destabilized (acute coronary pathology and/ or CVA in the last 6 months, serious asthma, serious heart failure, respiratory, lung or kidney failure, progressive inflammatory rheumatic disease…)
* Women under contraception and with a pregnancy project
* Patient already includes in a research protocol involving the human person
* Protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Decrease the impact of the fibromyalgia on the daily quality of life of the patients suffering of moderate fibromyalgia at 6 months by the practice of an adapted physical activity coupled with therapeutic education. | 6 months
  Evolution of the Fibromyalgia Impact Questionnaire (FIQ) at 6 months compared to baseline.

SECONDARY OUTCOMES:
Evaluation of the kinetic of the evolution at the inclusion, at short-term (3 months), at medium-term (6 months) and at long-term (12 months) of the FIQ (Fibromyalgia Impact Questionnaire). | 3, 6 and 12 months
  Evolution of the FIQ score between the inclusion, 3 months, 6 months and 12 months.
Compare the percentage of patients who achieve an FIQ<39 at 6 months (threshold defining an fibromyalgia impact weak). | 6 months
  Percentage comparison of the patients who achieve an FIQ<39 at 6 months.
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the hetero-evaluation by a doctor of the global health state.
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the self-assessment by the patient (Patient global assessment / Patient Global Impression of Change Scale).
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the Global Physical Activity Questionnaire (GPAQ)
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the Pain VAS
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the Pichot score (tiredness)
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the Questionnaire PSQI (Pittsburgh Sleep Quality Index).
Evaluate in a global way the disease evolution according to the 4 axis of the EULAR (pain, tiredness, sleep quality, physical activity). | 3, 6 and 12 months
  Evolution of fibromyalgia between the inclusion, 3 months, 6 months and 12 months according to the TSK (Tampa Scale for Kinesiophobia).
Improve the global quality of life | 3, 6 and 12 months
  Improvement of the questionnaire EQD-3L between the inclusion, 3 months, 6 months and 12 months.
Improve self-esteem | 3, 6 and 12 months
  Improvement of the score de Rosenberg between the inclusion, 3 months, 6 months and 12 months.
Improve the mood | 3, 6 and 12 months
  Improvement of the questionnaire HADS between the inclusion, 3 months, 6 months and 12 months.
Diminuate the health care consumption of the subjects at 3, 6 and 12 months compared to baseline. | 3, 6 and 12 months
  Decrease of the pharmacological consumption (by therapeutic class : analgesic, antidepressant, antiepileptic, other), medical and paramedical consultation, hospitalization, professional absenteeism, resort to complementary medicine between the inclusion, 3 months, 6 months and 12 months.
Improve the perception of the impact of the disease in the relations with close relations | 3, 6 and 12 months
  Evaluation by a close relation of the disease evolution and the relational impact via an VAS between the inclusion, 3 months, 6 months and 12 months.
Study the impact of the Fibrovelis program on the evolution of the muscular parameter. | 3 months (second to last trip of the intervention program).
  Change from baseline of the muscular parameters record by the Intelligent Electric Bike for the Health during an standardized stress test repeted at the end of after the intervention program.
Study the impact of the Fibrovelis program on the evolution of cardio-respiratory physiological efficiency parameter. | 3 months (second to last trip of the intervention program).
  Change from baseline of the cardio-respiratory physiological parameters record by the Intelligent Electric Bike for the Health during an standardized stress test repeted at the end of after the intervention program.
Evaluate the remanence of the long-term effect for the immediate intervention group | 18 months
  Evolution of the Fibromyalgia Impact Questionnaire (FIQ) and principal secondary outcomes at 18 months compared to Baseline for the immediate intervention group.
Evaluate the effect size of the intervention between 12 and 18 months for the diferred intervention group. | 12 and 18 months
  Evolution of the Fibromyalgia Impact Questionnaire (FIQ) and principal secondary outcomes at 18 months compared to 12 months for the diferred intervention group.
In the 2 groups, describe and analyze the effort adaptation in a population suffering of moderate fibromyalgia according the muscular power parameters. | 3 months
  Change from Baseline of the muscular power data.
In the 2 groups, describe and analyze the effort adaptation in a population suffering of moderate fibromyalgia according the cardio respiratory parameters. | 3 months
  Change from Baseline of the cardio respiratory physiological data.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Maindet, MD, Principal Investigator — University Hospital, Grenoble

REFERENCES:
- [Background] Wolfe F. Fibromyalgia: the clinical syndrome. Rheum Dis Clin North Am. 1989 Feb;15(1):1-18. PMID 2644671
- [Result] Cazzola M, Atzeni F, Salaffi F, Stisi S, Cassisi G, Sarzi-Puttini P. Which kind of exercise is best in fibromyalgia therapeutic programmes? A practical review. Clin Exp Rheumatol. 2010 Nov-Dec;28(6 Suppl 63):S117-24. Epub 2010 Dec 22. PMID 21176431
- [Result] Peterman JE, Morris KL, Kram R, Byrnes WC. Pedelecs as a physically active transportation mode. Eur J Appl Physiol. 2016 Aug;116(8):1565-73. doi: 10.1007/s00421-016-3408-9. Epub 2016 Jun 14. PMID 27299435
- [Result] Gojanovic B, Welker J, Iglesias K, Daucourt C, Gremion G. Electric bicycles as a new active transportation modality to promote health. Med Sci Sports Exerc. 2011 Nov;43(11):2204-10. doi: 10.1249/MSS.0b013e31821cbdc8. PMID 22005715
- See also: Gretchen Reynolds. The Surprising Health Benefits of an Electric Bike. July 6, 2016 6:00 AM July 6,2016 — https://well.blogs.nytimes.com/2016/07/06/the-surprising-health-benefits-of-an-electric-bike-2/